CLINICAL TRIAL: NCT01556516
Title: Pregnancy and Birth Outcome in Women With Pompe Disease
Status: Completed | Type: Observational
Sponsor: O & O Alpan LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 11-CFCT-02
Record Dates: First submitted 2012-03-09; First posted 2012-03-16 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with Pompe Disease

SUMMARY:
This study explores the outcome and effect of pregnancy on Pompe Disease. The results are expected to guide clinicians in counseling and care of women with Pompe disease, who are planning to become pregnant, and during the pregnancy.

DETAILED DESCRIPTION:
Pompe disease (glycogen storage disease type II) is a lysosomal storage disorder resulting from the deficiency of the enzyme acid alpha-glucosidase. Similar to many lysosomal storage diseases, the phenotypic spectrum in Pompe disease is varied, existing in infantile, and late-onset forms. In the classic infantile form, patients develop cardiomyopathy, resulting in premature death. In the later-onset forms, there is proximal muscle weakness similar to that of limb-girdle muscular dystrophy, which is associated with progressive weakness of different muscle groups. The primary morbidity in Pompe disease is associated with progressive respiratory insufficiency.

Events that act as metabolic stressors, in general, such as pregnancy may act as modifiers in lysosomal storage disorders. In much studied Gaucher disease, pregnancy increased the risk of acute bone crises, even in otherwise asymptomatic patients. However, similar studies lack for Pompe disease. Most data that is used to counsel patients with Pompe disease are derived from other muscular dystrophies, because obstetric risk and complications.

This is a retrospective case review study in female subjects age 18years and above. This study investigates the effects of acid alpha-glucosidase deficiency on pregnancy, pregnancy and disease outcomes in patients with adult-onset Pompe disease. The study will define the immediate effect of enzyme replacement therapy with Lumizyme/Myozyme on the outcomes of pregnancy and the fetus.

Subjects will be invited to participate through an initial mail or phone contact. If patient is interested, and agrees to participate in the study the study questionnaire will be provided to them. The patients then, need to complete the questionnaire, sign and date it and mail it back along with a release of any medical information forms. The returned signed and dated questionnaire from the patient serves as an indication of their consent to participate in the study. Alternatively, study PI or coordinator may review the questionnaire with the subject during a phone interview. However, the subject's signature is still required to attest to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Pompe disease
* Females age 18 and over
* Have been pregnant or anticipating pregnancy in near future.

Exclusion Criteria:

* If the diagnosis of Pompe disease is not confirmed
* If the subject is not able to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 female subjects (18 and above) who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Effect of pregnancy on Pompe disease severity and progression. | 5years
  The effect of pregnancy on Pompe disease severity and progression as measured by increase in muscle weakness, use of assistive devices for mobility or breathing based on subject's reporting.

SECONDARY OUTCOMES:
Effect of Pompe disease on pregnancy and pregnancy outcomes. | 5 years
  The effect of Pompe disease on pregnancy and pregnancy outcomes as measured by para-and peripartum complications, and fetal development based on subjects' reporting

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — O&O Alpan
Locations (1):
- O&O Alpan, Fairfax, Virginia, United States